CLINICAL TRIAL: NCT06746987
Title: The Effect of Theta Healing Meditation Technique Applied to Elderly Individulas on Sleep Quality and Psychological Well- Being
Brief Title: The Effect of Meditation Applied to Elderly Individulas on Sleep Quality and Psychological Well- Being
Acronym: Meditation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Nazmiye UĞUR, Mersin University Nursing PhD Student, Mersin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MersinUUU
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Sleep Quality and Psychological Well- Being
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental clinical trial with pre- test and post- test measurements consisting of a study and control group.
Masking Description: A single blind technique will be used in the research. Thus, it will not be known to the subjects whether the research participants are in the study or control groups. When the research is completed, the data of the study and control groups will be transferred to the computer environment by a researcher independent of the research, and the data will be analyzed by a statisitcian and the findings will ve reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meditation (Experimental): Study and control groups will be determined. Firstly, randomization of the study and control groups in the research will be done by an independent researcher on the randomizer.org website. Secondly, the Pitsburg Sleep Quality Scale and PERMA test will be applied to the study and control groups as a pre- test. Thirdly, theta healing meditation will be applied to the study group for 4 weeks, 2 days a week, 15- 30 minutes a day. After the 4 week meditation practice is completed with the study group, a final test will be given to the study and control groupsthe Pitsburg Sleep Quality Scale and PERMA test will be applied as the final test.
  Interventions: Other: Meditation

INTERVENTIONS:
Other: Meditation — After the appropriate sample group for the research is created, study and control groups will be determined. Firstly, randomization of the study and control groups in the research will be done by an independent researcher on the randomizer.org website. Secondly, the Pitsburg Sleep Quality Scale and PERMA test will be applied to the study and control groups as a pre- test. Thirdly, theta healing meditation will be applied to the study group for 4 weeks, 2 days a week, 15- 30 minutes a day. After the 4 week meditation practice is completed with the study group, a final test will be given to the study and control groupsthe Pitsburg Sleep Quality Scale and PERMA test will be applied as the final test.

SUMMARY:
It is planned as a randomized controlled experimental study to examine the effect of theta healing meditation technique on sleep quality and psychological well- being of elderly individuals.

DETAILED DESCRIPTION:
To evaluate the effect of theta healing meditation technique on sleep quality and psychological well- being in individuals over the age of 65, a study will be conducted with a total of 34 individuals consisting of a study and control group. Analysis of the research sample size was made using the G power 3.1.9.6 program. In the study, individuals who can communicate in Turkish, have received written and verbal permission to participate in the research, are over 65 years old, have a score of 24 or more on the Standardized Mini Mental Test (SMMT), have no preception disorder, and have no hearing problems will be included in the study. İndividuals who meet the research criteria for members of retirement homes will be included in the research. Sample selection will be completed in accordance with the study' s inclusion, axclusion criteria, followed by randomization. Individuals will be informed about the purpose of the research and the the research process, and the patient individuals will be given the ''Informed Voluntary Consent Form'' and ''Patient Introduction Form'', ''Pittsburg Sleep Quality Scale'' and ''Psychological Well- Being Scale (PERMA)'' as pre- tests, face to face, will be filled.Theta healing technique and meditation, visualization and thinking practice will be applied to the elderly individuals in the study group face to face under the guidance of the researcher for 20 minutes, 2 days a week, for 4 weeks.There will be no intervention in the control group for a 4 week period. After the 4- week theta healing meditation application is completed with the study group,''Pittsburg Sleep Quality Scale'' and ''Psychological Well- Being Scale (PERMA)'' scales will be applied to the study and control groups as a final test. The research will be competed by statistical analysis and reporting of the data obtained from the research.

ELIGIBILITY:
Inclusion Criteria:

* Written and verbal permission was obtained to participate in the research, Able to communicate in Turkish, Those aged 65 and over, Those who signed the informed consent form to participate in the research, Having a Standardized Mini Mental Test (SMMT) score of 24 points and above, No perception disorder, Without psychological medical diagnoses, Those without hearing problems will be included.

Exclusion Criteria:

* Standarzide Mini Mental Test (SMMT) score below 24 points, Having a perception disorder, Those with psychological medical diagnoses, Having hearing problems, Cannot communicate in Turkish, Those who have any health problems during the application process, Those who cannot continue the research for any reason, Those who want to leave the research with their own consent will not be included in the research.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-27 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
The effect of theta healing meditation on sleep quality will be evaluated with the Pittsburg Sleep Quality Scale. | The change before theta healing meditation and after 4 weeks of meditation lasting 15- 30 minutes, 2 days a week.
  The Pittsburg Sleep Quality, which examines the individual' s sleep quality in the last month, consists of 24 items. 24 items in the scale; It consists of 19 self- report questions answered by the individual and five questions answered or spouse and are not included and are not included in the scoring instructions and are used only for clinical information. Self- report questions included in the scoring consist of 7 components. These components; It provides information about subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency sleep disturbance, use of sleeping pills, and daytime sleep dysfunction. Each question is evaluated with a number from 0 to 3. The highest score that can be obtained from the scale is 21. An increase in the score obtained from the scale indicates that sleep quality is poor.

SECONDARY OUTCOMES:
The effect of theta healing meditation on psychological well- being will be evaluated with the Psychological Well- Being Scale. | The change before theta healing meditation and after 4 weeks of meditation lasting 15- 30 minutes, 2 days a week.
  Psychological Well- Being Scale five dimensions include positive emotions, positive emotions, positive relationships, meaning, achievement and connection. It is found bu taking the average.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes